CLINICAL TRIAL: NCT02516397
Title: Randomised Controlled Trial, Double-blind, to Measure Efficiency and Tolerance of a New Food Supplement OMNIA on Body Fat Mass Reduction in Overweight Subjects
Brief Title: OMNIA Efficacy on Body Fat Mass Reduction
Acronym: PEPOLUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated because of conflicting results from intermediate analysis.
Sponsor: Vivatech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID : 2014 -A01889-38
Record Dates: First submitted 2015-07-28; First posted 2015-08-05 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Overweight
Keywords: body fat mass reduction
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omnia group (Experimental): After 2 weeks of run-in period, subjects take 2 Omnia pills per meal (3 meals a day) for 12 weeks.
  Interventions: Dietary Supplement: Omnia
- Placebo group (Placebo Comparator): After 2 weeks of run-in period, subjects take 2 Placebo pills per meal (3 meals a day) for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omnia — 12weeks of treatment
  Arms: Omnia group
Dietary Supplement: Placebo — 12weeks of treatment
  Arms: Placebo group

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of a food supplement OMNIA compared to a placebo in reducing the body fat mass in 70 overweight subjects during 12 weeks treatment.

DETAILED DESCRIPTION:
Overweight and obesity represent a serious public health issue. These conditions are characterized by an abnormal or excessive accumulation of body fat mass and they are related to an increase risk of developing chronic diseases such as cardiovascular, diabetes, arthrosis and certain kind of cancer (breast; colon). It's thus necessary to find new products able to counteract both overweight and obesity.

Omnia is a food supplement based on a Phaseolus vulgaris extract. It has pancreatic amylase inhibition properties.

In the following clinical trial, OMNIA will be administrated to a group of overweight subjects in order to evaluate its efficacy on reducing the body fat mass. Its action will be compared to a placebo administered to a second group of overweight volunteers with the same modalities as OMNIA.

ELIGIBILITY:
Inclusion Criteria:

* 25≤ BMI<30 kg/m2
* excess of fat mass
* food habits : 3 meals a day and a glucides intake equivalent to at least 40% of daily energy (i.e.: glucides intake at each meal)
* Able to give a written or verbal informed consent
* Affiliated or beneficiary of social security

Exclusion Criteria:

* Weight loss/gain > 2kg within the preselection period (2 weeks)
* Abnormal blood results at V0
* Physical activity (sport; lifestyle) modification planned or ongoing during the trial
* Severe pathologies/disorders (bulimia; anorexia; diabetes; cancer…) emerging
* Pregnancy during the study
* Consent withdrawal
* Allergy to Omnia
* observance <60%
* Investigator or promotor decision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Reduction of body fat mass loss measured by DEXA (Dual-energy X-ray absorptiometry) | 12 weeks

SECONDARY OUTCOMES:
change from baseline in Body Mass Index (BMI) | 6, 12 weeks
change from baseline on the ratio fat/lean body mass measured by DEXA | 12 weeks
change from baseline on weight | 6, 12 weeks